CLINICAL TRIAL: NCT02666222
Title: To Evaluate the Long-term Safety and Efficacy of the Esteem® Hearing Implant in Subjects Suffering From Moderate to Severe Hearing Loss
Brief Title: The Esteem® Hearing Implant Post Approval Study
Status: Completed | Type: Observational
Sponsor: Envoy Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 0204 Post-Approval Study (PAS)
Record Dates: First submitted 2011-07-08; First posted 2016-01-28 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-01

CONDITIONS: Hearing Loss
Keywords: hearing loss; sensorineural; hearing implant
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: The Esteem Hearing Implant — The Esteem® Hearing Implant is designed to improve hearing in subjects suffering from moderate to severe hearing loss that is sensorineural in origin. The Esteem® has been approved by FDA for the US market under Pre-Market Approval P090018 and this study fulfills the requirement for one of the Post Approval Studies.

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of the Esteem® Hearing Implant in subjects suffering from moderate to severe hearing loss.

DETAILED DESCRIPTION:
The Post Approval Study is an extension of the pivotal clinical trial, which was designed as a prospective, multi-center, non-randomized, clinical trial to evaluate the safety and efficacy of the Esteem® System. For this trial the subject acts as his or her own control.

This trial has been designed to meet the United States' regulatory requirements.

The subjects included in this study include the 57 subjects implanted under the original Investigational Device Exemption (IDE) study and the five (5) subjects implanted under the continued access expansion approved by the FDA. Of these 62 subjects, all but one (explant) were available for continued follow-up. These subjects were re-consented for the 5 year Post Approval Study. No new subjects were enrolled and implanted in this study. The goal was to monitor a minimum of 45 subjects through their five (5) year follow-up. Ultimately, 51 subjects completed the study.

The following questions are to be answered:

* Is the Esteem effective through 5 year follow-up?
* Is the Esteem safe through 5 year follow-up?

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following criteria to be eligible for treatment in the trial:

1. Subject is at least 18 years old
2. Subject understands the nature of the procedure and has signed the Subject Informed Consent Form prior to the procedure
3. Subject is willing and able to comply with specified follow-up evaluations and understands the audiological test procedures and use of the Esteem® System.
4. Subject has moderate to severe sensorineural hearing loss between 500 and 4000 Hz in the ear to be implanted with pure tone air-conduction threshold levels within the limits of a Hearing Aid (HA) as follow:

   Freq (Hz) 500 1000 2000 3000 4000 Lower Level (dB HL) 30 35 35 35 35 Upper Level (dB HL) 100 100 100 100 100
5. Subject's air-bone gap is no greater than 10 dB at 4 of the 5 following frequencies: 500, 1000, 2000, 3000 and 4000 Hz.
6. Subject has an unaided maximum word recognition score of greater than or equal to 40% with recorded delivery using a phonetically balanced word list at Speech Reception Threshold (SRT) + 40 dB or at maximum tolerable presentation level.
7. Subject is a current user of a properly functioning and appropriately fit hearing aid. This is defined as the subject has used this aid for at least four (4) hours (average) per day (in the ear to be implanted) for at least three (3) months for a new aid or one (1) month for an adjusted aid.
8. Subject's hearing aid, in the ear to be implanted, shall appropriately fit optimally.
9. Subject has normally functioning eustachian tube
10. Subject has normal tympanic membrane
11. Subject has a normal middle ear anatomy
12. Subject has adequate space for Esteem® System implant determined via fine cut temporal bone CT scan
13. Subject is a native speaker of the English language.
14. Subject is a hearing aid user in the ear to be implanted

Exclusion Criteria:

Subjects will be excluded from the trial if any one of the following criteria is met:

1. Subject has a history of post-adolescent chronic middle ear infections, inner ear disorders or recurring vertigo requiring treatment, disorders such as mastoiditis, Hydrops or Meniere's syndrome or disease
2. Subject has a history of external otitis or eczema for the outer ear canal and the investigator believes this will affect the Esteem® System implantation
3. Subject has cholesteatoma or destructive middle ear disease
4. Subject has life expectancy of less than two (2) years due to other medical conditions
5. Subject has retrocochlear or central auditory disorders
6. Subject is known to be suffering from any psychological, developmental, physical, or emotional disorder that the investigator feels would interfere with the surgery or follow-up testing
7. Subject has a known history of fluctuating air conduction and/or bone conduction hearing loss over a one-year period of 15 dB in either direction at 2 or more frequencies (from 500 - 4000 Hz)
8. Subject has sudden hearing loss due to unknown cause
9. Subject has a history of disabling tinnitus, defined as tinnitus which required treatment.
10. Subject is unable to adequately perform audiological testing
11. Subject has a medical condition or undergoing a treatment that may affect healing and the investigator does not believe the subject is a good candidate for the trial.
12. Subject has diabetes that is not well controlled with medication or diet and the investigator does not believe in his best medical judgment that the subject would be a good candidate for the trial
13. Subject is pregnant at the time of device implant
14. Subject has a history of keloid formation
15. Subject has known hypersensitivity to silicone rubber, polyurethane, stainless steel, titanium and/or gold

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons suffering from moderate to severe hearing loss that is sensorineural in origin
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2010-08; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Shohet, MD, Principal Investigator — Hoag Memorial Hospital; Elizabeth H Toh, MBBS; MD, Principal Investigator — Lahey Clinic Medical Center; Eric M Kraus, MD, MS, FACS, Principal Investigator — Moses H. Cone Memorial Hospital
Locations (5):
- United States (5):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Shohet Ear Associates, Newport Beach, California
  - Lahey Clinic, Inc., Burlington, Massachusetts
  - Surgical Care Affiliates, Greensboro, North Carolina
  - The Ear Center of Greensboro, Greensboro, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Invisible Hearing with Esteem® — http://www.envoymedical.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- Esteem Implant: Subjects implanted with the Esteem Totally Implantable Hearing System
Period: Overall Study
Arm/Group | Esteem Implant
Started | 51
Completed | 49
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Esteem Implant
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 34
Race/Ethnicity, Customized [Number; unit: participants]
  White/Caucasian | 50
  Black/Non-Hispanic | 0
  Hispanic | 0
  Asian | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Pre-implant Aided Condition) at Year 5 in Speech Reception Threshold (SRT)
Description: ENDPOINT #1: SRT at baseline minus SRT at Year 5. Positive difference (i.e. lower value of SRT with the Esteem) indicates better outcome.
Time Frame: Baseline through Year 5 of Follow Up
Population: 5 Year Follow-up
Measure: Mean (Standard Error); unit: dB
Arm/Group | Esteem Implant
Number analyzed (Participants) | 49
dB | 4.8 (2)

2. Primary Outcome: Change From Baseline (Pre-implant Aided Condition) at Year 5 in Word Recognition Score (WRS) at 50 dB HL
Description: ENDPOINT #2: WRS at Year 5 minus WRS at baseline. Positive difference (in % correct) indicates better outcome.
Time Frame: Baseline through Year 5 of Follow Up
Population: 5 Year Follow-up Visit
Measure: Mean (Standard Error); unit: percentage of correct responses
Arm/Group | Esteem Implant
Number analyzed (Participants) | 49
percentage of correct responses | 17 (4.2)

3. Primary Outcome: Incidence of Serious Adverse Device Events (SADEs) and Device Failures and Replacements at Each Follow-up.
Description: ENDPOINT #3: The analysis of the incidence of SADEs and device failures and replacements at each follow-up.
Time Frame: SADEs, PAS phase through Year 5 of Follow Up
Population: Cumulative through 5-Year Follow-up
Measure: Number; unit: participants
Arm/Group | Esteem Implant
Number analyzed (Participants) | 51
participants | 3

4. Primary Outcome: Bone Conduction Stability
Description: ENDPOINT #5: Difference between Baseline and 5 Year Pure-Tone Average (PTA; average of 500, 1000, 2000 Hz thresholds); calculated as PTA at Year 5 minus PTA at baseline. Smaller magnitude dB difference indicates better outcome.
Time Frame: Baseline through 5 Year Follow-Up
Population: Difference between Baseline and 5 Year PTA (average of 500, 1000, 2000 Hz thresholds)
Measure: Mean (Standard Error); unit: dB
Arm/Group | Esteem Implant
Number analyzed (Participants) | 49
dB | 3.7 (1.1)

5. Secondary Outcome: Improvement in Quality of Life as Reflected by Abbreviated Profile of Hearing Aid Benefit (APHAB) Questionnaire
Description: APHAB results were obtained from baseline aided condition through Year 5 of follow up. The APHAB responses are in terms of percent of time an individual experiences problems, on a scale of 0-100%; lower scores indicate fewer problems.Compared scores with Esteem to scores in baseline aided condition, calculated as APHAB Global score at baseline minus APHAB Global score at Year 5, giving a "difference in benefit" score. The Global Score is the mean of the scores (% of problems) for Ease of Communication (EC), Reverberation (RV), and Background Noise (BN) subscales of the APHAB. A positive difference in benefit score indicates more benefit with Esteem.
Time Frame: Baseline through Year 5 of Follow Up
Population: 5 Year Follow-up
Measure: Mean (Full Range); unit: difference score in units on a scale
Arm/Group | Esteem Implant
Number analyzed (Participants) | 47
difference score in units on a scale | 5.6 [.4 to 10.9]

ADVERSE EVENTS:
Time Frame: PAS phase through 5 years
Description: All Adverse Events adjudicated by Clinical Events Committee
Arm/Group | Esteem Implant
Serious Adverse Events (participants affected / at risk) | 14/51
Other Adverse Events (participants affected / at risk) | 42/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esteem Implant (N=51)
Sore behind ear (Skin and subcutaneous tissue disorders) | 1 (1)
Exposed Leads (General disorders) | 1 (1) — Post-auricular area
Infected Implant Site (Infections and infestations) | 1 (1)
Gall bladder removal surgery (Gastrointestinal disorders) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 1 (1)
Cancer treatment (Surgical and medical procedures) | 1 (1)
Disc displacement (Musculoskeletal and connective tissue disorders) | 1 (1)
Fell and broke collarbone, clavicle & 3 ribs. Slight lung puncture. (Injury, poisoning and procedural complications) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Shoulder surgery (Surgical and medical procedures) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Death (Social circumstances) | 2 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Esteem Implant (N=51)
Distortion (Ear and labyrinth disorders) | 1 (1)
Facial Tingling and Weakness (Nervous system disorders) | 1 (1)
Feedback (General disorders) | 1 (1)
Incision Site Pain/Soreness (Skin and subcutaneous tissue disorders) | 2 (2)
Low Performance (Ear and labyrinth disorders) | 1 (1)
Mild Discomfort at Processor Site (Skin and subcutaneous tissue disorders) | 1 (1)
Pain Around Processor Ridge (Skin and subcutaneous tissue disorders) | 1 (1)
Positional Vertigo (Ear and labyrinth disorders) | 1 (1)
Postauricular skin "shrink-wrapped" around leads (Skin and subcutaneous tissue disorders) | 1 (1)
Tenderness and drainage at incision site (Skin and subcutaneous tissue disorders) | 1 (1)
Neck pain (General disorders) | 1 (1)
Poorly performing implant (Ear and labyrinth disorders) | 1 (1)
Premature battery depletion (General disorders) | 1 (1)
Reduced performance (Ear and labyrinth disorders) | 1 (1) — Reduced SRT/PTA functional gain
Abscess left external auditory canal (Ear and labyrinth disorders) | 1 (1)
Ear infection, both ears (Ear and labyrinth disorders) | 1 (1)
Eyelid lift; both eyes (Surgical and medical procedures) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
High blood pressure (Cardiac disorders) | 1 (1)
Impacted cerumen, right ear (Ear and labyrinth disorders) | 1 (1)
Low platelets (Blood and lymphatic system disorders) | 1 (1)
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 (1)
Sinus infection (Infections and infestations) | 1 (1)
Sinus symptoms, cold (Infections and infestations) | 1 (1)
Strep throat, resolving (Infections and infestations) | 1 (1)
Tympanic membrane hematoma (Ear and labyrinth disorders) | 1 (1) — with minor flame hemorrhage
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Arthritis, R shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Brown's syndrome (Eye disorders) | 1 (1)
Cataract surgery (Eye disorders) | 1 (1)
Enlarged prostate (Renal and urinary disorders) | 1 (1)
Knee replacement (Surgical and medical procedures) | 1 (1)
Loss of balance (Ear and labyrinth disorders) | 1 (1)
Otitis Externa (Ear and labyrinth disorders) | 1 (1)
Sacroiliitis (Infections and infestations) | 1 (1)
Sinus congestion, sinus disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
TIA (Cardiac disorders) | 1 (1)
Increased tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo vs. disequilibrium (Ear and labyrinth disorders) | 1 (1)
Pain (Ear and labyrinth disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
1. Study endpoints do not account for natural progression of hearing loss over 5-year follow-up.
2. Fitting methods for pre-implant hearing aid were not strictly controlled in the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less